CLINICAL TRIAL: NCT06718283
Title: Assessment of Hematologic Indices in Juvenile Lupus Erythematosus Patients : Correlation With Disease Activity and Chronic Organ Damage in These Patients
Brief Title: Assessment of Hematologic Indices in Juvenile Lupus Erythematosus Patients:Correlation With Disease Activity and Chronic Organ Damage in These Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alshimaa Hamdey Khalaf, Assistant lecturer- Rheumatology and Rehabilitation department, Sohag University
Other Study IDs: Soh-Med-24-11_3MD
Record Dates: First submitted 2024-11-25; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Systemic Lupus Erythematosus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim to evaluate the relationship between some important hematologic indices in juvenile lupus erythematosus patients and if these indices may be use as markers of disease acitivity in these patients or not ,also evaluate the relationship with these markers and chronic organ damage index

DETAILED DESCRIPTION:
We calculate important hematologic indices in children diagnosed as SLE as systemic inflamatory index ,systemic inflamatory response index and aggregate index of systemic inflamation in these patients ,and correlate these indices with SLE disease activity index and chronic damage index in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who fillful 2012 SLICC criteria or 2019 ACR/EULAR criteria of systemic lupus erythematosus
* Age of patients at disease onset before 18 years

Exclusion Criteria:

* Adult onset disease ( age at disease onset after 18 years
* Any other chronic inflamatory disorders or other autoimmune diseases

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients males or females below age of 18 years diagnosed as juvenile systemic lupus erythematosus based on 2012 SLICC criteria or 2019 ACR/EULAR criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Calculation of hematological indices in juvenile lupus erythematosus patients | 3_ 6 months
  Calculation of systemic inflamatory index,systemic information response index and aggregate index of systemic inflamation ,and correlate these indices to SLE disease activity index
Correlation between hematologic indices in juvenile lupus erythematosus patients and disease activity in these patients | 3-6 months
  SLEDAI score in juvenile lupus erythematosus patients

SECONDARY OUTCOMES:
Calculation of chronic damage index in juvenile lupus erythematosus patients | 3_6 months
  SLICC/ACR score in juvenile lupus erythematosus patients
Relationship between hematologic index and chronic organ damage index in juvenile lupus erythematosus patients | 3-6 months
  SLICC/ACR score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aringer M, Petri M. New classification criteria for systemic lupus erythematosus. Curr Opin Rheumatol. 2020 Nov;32(6):590-596. doi: 10.1097/BOR.0000000000000740. PMID 32925250
- [Background] Liu P, Li P, Peng Z, Xiang Y, Xia C, Wu J, Yang B, He Z. Predictive value of the neutrophil-to-lymphocyte ratio, monocyte-to-lymphocyte ratio, platelet-to-neutrophil ratio, and neutrophil-to-monocyte ratio in lupus nephritis. Lupus. 2020 Aug;29(9):1031-1039. doi: 10.1177/0961203320929753. Epub 2020 Jun 5. PMID 32501169
- [Background] Hassan MR, Hossain A, Mahata J, Srivastava V, Sarkar S. Hematological manifestation of Pediatric Systemic Lupus Erythematosus (SLE) - A single centered cross-sectional study. J Family Med Prim Care. 2024 May;13(5):1787-1792. doi: 10.4103/jfmpc.jfmpc_1583_23. Epub 2024 May 24. PMID 38948621